CLINICAL TRIAL: NCT05704803
Title: Prospective, Multi-Center, Non-Randomized Study to Evaluate OTC At Home SARS-CoV-2 Molecular Diagnostic Test
Brief Title: COVID-19 Molecular OTC At Home Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3EO Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3EO-CoV2-02
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study Groups (Experimental): Positives: Symptomatic vs. Asymptomatic Negatives: Symptomatic vs. Asymptomatic
  Each broken down by age groups:
  2-14 years old 15-24 years old 25-64 years old 65+ years old
  Interventions: Diagnostic Test: Diagnostic Test: IN Vitro

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: IN Vitro — In vitro diagnostic test for COVID-19 using anterior nasal swabs.

SUMMARY:
The objective of this study is to evaluate the a molecular, OTC/At-Home COVID-19 Test in individuals presenting at a medical facility. In eligible subjects, nasal samples will be collected for use with the at-home molecular COVID-19 Test, which will be compared to the Zymo® rRT-PCR test results obtained via samples specified by the sponsor (e.g., AN [anterior nares] swab) to determine accuracy of the at-home/OTC molecular COVID-19 Test in detecting COVID-19 in participants.

DETAILED DESCRIPTION:
The molevular, at-home COVID-19 Test is a unique rapid molecular test system intended to detect SARS-CoV-2 virus in the OTC setting using a dedicated reusable test reader to test nasal swab samples. Early testing will help to determine limit of detection (LOD) of the molecular COVID-19 Test and will be compared to a sensitive molecular test that has been authorized for emergency use by the FDA. The COVID-19 Test will leverage the processing and testing of the associated Swab device when inserted directly into the reaction tube (Key) where reverse transcription, Loop-Mediated Isothermal DNA Amplifications (LAMP) processing and sequence-specific probe technologies to detect segments of the SARS-CoV-2 genome are managed automatically by the reusable test reader.

ELIGIBILITY:
All Participants must meet ALL of the following:

1. ≥ 2 years of age. Subjects ages 2 ≤ x ≤ 17 will provide assent in addition to parent / legal guardian's consent.
2. Able to read and write in English and/or Spanish (subjects or guardians)
3. Willing and able to provide informed consent (subject or Legally authorized Representative (LAR)). Subjects unable to consent will provide assent in addition to LAR consent.

Symptomatic Participants must meet BOTH of the following:

1. Have at least one of the following symptoms the day of the test:

   1. Fever
   2. Cough
   3. Shortness of Breath
   4. Difficulty Breathing
   5. Muscle Pain
   6. Headache
   7. Sore Throat
   8. Chills
   9. New loss of taste or smell
   10. Congestion
   11. Runny nose
2. Onset of symptoms occurred within the past 7 calendar days.

Asymptomatic Participants must meet BOTH of the following:

1. Not experiencing any of the following symptoms at the time of specimen collection and testing: fever, cough, shortness of breath or difficulty breathing, new loss of taste or smell, muscle or body aches, headache, sore throat, congestion or runny nose, nausea or vomiting or diarrhea.
2. Exposed to known COVID-19 positive individuals or are suspected to have had COVID-19 over the past 7 calendar days.

Exclusion Criteria:

Participants must not meet ANY of the following:

1. Eating or drinking 30 minutes prior, or smoking 60 minutes prior to specimen collection.
2. Unable to tolerate sample collection, or has contraindications to collection such as nasal bleeding, ulcers, or surgery within the past 3 months.
3. Underwent a nasal wash / aspirate as part of standard of care < 24 hours prior to the study start.
4. Currently receiving or has received within the past 30 days of the study visit an experimental drug, biologic, or device including treatment or therapy.
5. Previously participated in this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Correlation of the 3EO Health SARS-CoV-2 standard of care (PCR) Zymo rRT-PCR results of the anterior nare sample. | 1-16 weeks
  The primary endpoints of this study will be the correlation of the 3EO Health SARS-CoV-2 OTC At Home Test results from nasal samples to the comparator, standard of care (PCR) Zymo rRT-PCR results of the anterior nare sample

CONTACTS AND LOCATIONS:
Overall Officials: Adelina Paunescu, PhD, Study Director — Medicept Inc.
Locations (4):
- United States (4):
  - Bright Research Center, Miami, Florida
  - I.V.A.M. Clinical & Investigational Center, Miami, Florida
  - Vytalus Medical Atascocita, Humble, Texas
  - Vytalus Medical, Kingwood, Texas

IPD SHARING:
Plan to Share IPD: No